CLINICAL TRIAL: NCT01688453
Title: Reduction of Inequalities in Overweight and Obesity Management Care Access Among High School Adolescents
Brief Title: Overweight Management and Social Inequalities
Acronym: PRALIMAP-INES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: C11-46
Record Dates: First submitted 2012-09-07; First posted 2012-09-19 (Estimated); Last update posted 2025-12-10 (Actual); Status verified 2021-08

CONDITIONS: Overweight
Keywords: overweight/obesity; adolescence; care management
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1: (Active Comparator): Socially advantaged overweight or obese adolescents are allocated to the standard care management.
  Interventions: Behavioral: Standard care management
- Group 2 (Experimental): Socially less advantaged overweight or obese adolescents are allocated to the standard care management.
  Interventions: Behavioral: Standard care management
- Group 3 (Experimental): Socially less advantaged overweight or obese adolescents are allocated to the strengthened care management.
  Interventions: Behavioral: The strengthened care management

INTERVENTIONS:
Behavioral: Standard care management — The standard-care management program consists of 5 collective sessions of 2 hr each about nutritional practices (food and physical activity) and on changes of nutritional behaviours. The sessions are organized in high schools by the healthcare team in collaboration with pediatricians, dietitians and the Sickness Insurance Primary Fund.
  Arms: Group 1:; Group 2
Behavioral: The strengthened care management — The strengthened care management is the addition of the standard care management and of additional interventions.
  The standard-care management program consists of 5 collective sessions of 2 hr each about nutritional practices (food and physical activity) and on changes of nutritional behaviours. The sessions are organized in high schools by the healthcare team in collaboration with pediatricians, dietitians and the Sickness Insurance Primary Fund.
  The additional interventions are strengthened solicitation and accompaniment, peer-led education, motivational interview, financial support for physical activity practice, cooking classes and meetings of multidisciplinary consultation.
  Arms: Group 3

SUMMARY:
Background: The prevalence of overweight and obesity continues to increase in socially less advantaged populations but is stabilizing even is decreasing in socially more advantaged populations. The PRALIMAP trial highlighted the effectiveness of structured screening and care management in decreasing the prevalence of overweight and obesity in high school adolescents over 2 years. The PRALIMAP-INES trial aims to investigate whether a strengthened care management (CM) for socially less advantaged adolescents in school in the short and long term has an equivalent effect as a standard-CM on decreasing the prevalence of overweight and obesity among socially advantaged adolescents.

Intervention: PRALIMAP-INÉS is a mixed prospective and multicenter trial of 1,250 overweight and obese adolescents aged 13 to 18 years who are attending grade 9 and 10 in the 35 state-run schools of the Vosges department (northeastern France) for the academic years 2012-2013 2013-2014 and 2014-2015. Overweight adolescents (including obese) classified as advantaged are allocated to the standard-CM and those less advantaged are randomized to standard CM or strengthened-CM. The standard-CM consists of 5 collective sessions of 2 hr each performed in high school and supervised by a healthcare mobile team specialised in overweight and obesity care management for adolescents. The strengthened-CM consists of 5 collective sessions with the same standard operating procedure as the standard-CM with supplementary interventions between each session: strengthened solicitation with the adolescent and the family, peer-led educational sessions, motivational interviews, financial support for physical activity practice, cooking classes and multidisciplinary consultation meetings. Data on sociodemographics, anthropometrics, physical activity and mental health are collected at 3 visits: at the entry to grade 9 or 10 (before the intervention=T0), at the end of grade 9 or 10 (at the end of the intervention=T1) and at the end of grade 11 (1 year after the intervention=T2). Process evaluation data are also collected during the trial.

Expected results: To confirm the effectiveness of overweight CM for adolescents in a school setting and to highlight or not the effectiveness of specific strengthened interventions adapted for socially less advantaged adolescents to maintain social equality in access to overweight care.

DETAILED DESCRIPTION:
Background: The prevalence of overweight and obesity continues to increase in socially less advantaged populations but is stabilizing even is decreasing in socially more advantaged populations. The PRALIMAP trial confirmed major social inequalities in overweight and obesity frequency in adolescents in grade 10. The trial highlighted the effectiveness of structured screening and care management in decreasing the prevalence of overweight and obesity in high school adolescents over 2 years. The PRALIMAP-INES trial aims to investigate whether a strengthened care management strategy for socially less advantaged adolescents in school in the short and long term (just after the intervention and 1 year later) has an equivalent effect as a standard-care management strategy on decreasing the prevalence of overweight and obesity among socially advantaged adolescents.

Hypothesis: A strengthened overweight and obesity care management strategy for overweight and obesity (risk factors of cancer) can improve care access for socially less advantaged adolescents and maintain social equality in terms of overweight and obesity prevalence.

Intervention: PRALIMAP-INÉS is a mixed prospective and multicenter trial (one randomised part and one non-randomised part) of 1,250 overweight and obese adolescents aged 13 to 18 years who are attending grade 9 and 10 in the 35 state-run schools of the Vosges department (northeastern France) for the academic years 2012-2013, 2013-2014 and 2014-2015. After a session to detect overweight and obese adolescents, the social status of included adolescents as "advantaged" or "less advantaged" is determined. Adolescents classified as advantaged are allocated to the standard-care management and those less advantaged are randomized to standard-care management or strengthened-care management. The standard-care management consists of 5 collective sessions of 2 hr each performed in high school and supervised by a healthcare mobile team specialised in overweight and obesity care management for adolescents. The team consists of physicians, dietitians, psychologists and sports educators from the AVRS Association. The content of sessions was validated in the PRALIMAP trial. The strengthened-care management consists of 5 collective sessions with the same standard operating procedure as the standard-care management with supplementary interventions between each session: strengthened solicitation with the adolescent and the family, peer-led educational sessions, motivational interviews, financial support for physical activity practice, cooking classes and multidisciplinary consultation meetings (adjusting the care management according to the social status). Data on sociodemographics, anthropometrics, physical activity and mental health are collected at 3 visits: at the entry to grade 9 or 10 (before the intervention = T0), at the end of grade 9 or 10 (at the end of the intervention = T1) and at the end of grade 10 or 11 (1 year after the intervention = T2). T1 measurement allows for evaluating the short-term effect of the intervention and T2, the long-term effect of a 1-year break from the intervention. Data on participation and from questionnaires, as well as focus group and activity reports, necessary for evaluation, are collected during the trial.

Expected results: With this trial, the investigators expect to confirm the effectiveness of overweight and obesity care management for adolescents in a school setting and to highlight or not the effectiveness of specific strengthened interventions adapted for socially less advantaged adolescents to maintain social equality in access to overweight and obesity care.

ELIGIBILITY:
Inclusion criteria

* Attending grade 9 or 10 in one of the 35 state-run school of the Vosges department and be in a general, technological or vocational course,
* Aged ≤ 18 years old,
* not giving written refusal to participate in the trial,
* able to complete a questionnaire,
* overweight or obese according to the IOTF criteria (for BMI) and the McCarthy criteria (for waist circumference) and/or have a high eating disorder score, and/or express the need for management of excess weight,
* confirmed as corresponding to the 4 previous inclusion criteria by the physician, with elimination of adolescents with false-positive BMI (particularly athletic adolescents),
* agree to an overweight and obesity care management program.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1689 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Change in Body Mass Index from to baseline to 1 and 2 years | 0-1-2 years
  BMI is measured at baseline(on grade 10 entry) and after 1 and 2 follow up years(at the end of grades 10 and 11).
Change in overweight and obesity status according to IOTF norms | up to 2 years
  overweight and obesity status is calculated from BMI at each measurement time according to the IOTF norms for age and sex
Change in BMI Z score from baseline to one and two years | up to 2 years
  BMI Z score is calculated from BMI at each time measurement using WHO reference and SAS macro

SECONDARY OUTCOMES:
Change in waist circumference | 2 years
  waist circumference is measured two times at each measurement point by trained nurses and validated by a practitioner
change in eating attitude score from baseline to 1 and 2 years | up to 2 years
  Eating attitudes are measured at each measurement point using then EAT40 questionnaire
Change in anxiety and depression scores from baseline to 1 and 2 years | up to 2 years
  HAD questionnaire is used to measure score at each follow-up point

OTHER OUTCOMES:
Change in Nutritional behavior from baseline to 1 and 2 years | up to 2 years
  Nutritional behavior is measured through self administered questionnaires which allow to assess the compliance to French national recommendations

CONTACTS AND LOCATIONS:
Overall Officials: Serge Briançon, Pr, Principal Investigator — University of Lorraine
Locations (1):
- School, Nancy, Vosges, France

REFERENCES:
- [Result] Saez L, Langlois J, Legrand K, Quinet MH, Lecomte E, Omorou AY, Briancon S; PRALIMAP-INES Trial Group. Reach and Acceptability of a Mobile Reminder Strategy and Facebook Group Intervention for Weight Management in Less Advantaged Adolescents: Insights From the PRALIMAP-INES Trial. JMIR Mhealth Uhealth. 2018 May 18;6(5):e110. doi: 10.2196/mhealth.7657. PMID 29776897
- [Result] Saez L, Legrand K, Alleyrat C, Ramisasoa S, Langlois J, Muller L, Omorou AY, De Lavenne R, Kivits J, Lecomte E, Briancon S; PRALIMAP-INES Trial Group. Using facilitator-receiver peer dyads matched according to socioeconomic status to promote behaviour change in overweight adolescents: a feasibility study. BMJ Open. 2018 Jun 22;8(6):e019731. doi: 10.1136/bmjopen-2017-019731. PMID 29934380
- [Result] Legrand K, Lecomte E, Langlois J, Muller L, Saez L, Quinet MH, Bohme P, Spitz E, Omorou AY, Briancon S; PRALIMAP-INES trial group. Reducing social inequalities in access to overweight and obesity care management for adolescents: The PRALIMAP-INES trial protocol and inclusion data analysis. Contemp Clin Trials Commun. 2017 Jun 16;7:141-157. doi: 10.1016/j.conctc.2017.05.010. eCollection 2017 Sep. PMID 29696179
- [Result] Manneville F, Omorou AY, Legrand K, Lecomte E, Rydberg JA, Briancon S, Guillemin F; PRALIMAP Trial Group. Sociodemographic and psychological characteristics associated with discrepancy between body satisfaction and weight change among adolescents. Prev Med. 2021 Sep;150:106668. doi: 10.1016/j.ypmed.2021.106668. Epub 2021 Jun 1. PMID 34087324
- [Result] Omorou AY, Manneville F, Langlois J, Legrand K, Bohme P, Muller L, Guillemin F, Briancon S, Lecomte E; PRALIMAP-INES Trial Group. Physical activity rather than sedentary behaviour is socially determined in French adolescents with overweight and obesity. Prev Med. 2020 May;134:106043. doi: 10.1016/j.ypmed.2020.106043. Epub 2020 Feb 22. PMID 32097754
- [Derived] Dakin M, Manneville F, Langlois J, Briancon S, Lecomte E, Spitz E, Legrand K, Bohme P, Guillemin F, Omorou A. Role of dietary intake and physical activity in reducing weight social inequalities among adolescents: an application of G-formula to PRALIMAP-INES trial. Br J Nutr. 2024 Jul 28;132(2):182-191. doi: 10.1017/S0007114524001090. Epub 2024 May 27. PMID 38800976
- [Derived] Julia C, Omorou A, Lecomte E, Langlois J, Touvier M, Hercberg S, Briancon S, Kesse-Guyot E, Guillemin F; PRALIMAP-INES Trial Group. Behavioural risk patterns in adolescents with excess weight participating in the PRALIMAP-INES trial. Public Health Nutr. 2023 Jan;26(1):96-105. doi: 10.1017/S136898002200057X. Epub 2022 Mar 11. PMID 35272723